CLINICAL TRIAL: NCT01152931
Title: Antioxidant Micronutrients in Malaria:a Randomised Clinical Trial
Brief Title: Antioxidant Micronutrients in Malaria
Acronym: AMM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Lagos, Nigeria (Other)
Responsible Party: Dr Iribhogbe Osede Ignis, Department of Pharmacology and Therapeutics, College of Medicine Ambrose Alli University, Ekpoma.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULagosclinicaltrials; ULCT123456 (Registry Identifier: ULCT123456); ULCT123456 (Registry Identifier: Ministry of Health); HCC8/T2A/443111 (Registry Identifier: HCC8/T2A/443)
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2010-08

CONDITIONS: Malaria
Keywords: Antioxidants; Micronutrients; Malaria; focus is to determine the effect of antioxidant micronutrients in malaria
MeSH Terms: conditions — Malaria | interventions — amodiaquine, artesunate drug combination; Artemether, Lumefantrine Drug Combination; Artesunate; Vitamin A; Vitamin E; Zinc; Selenium; Amodiaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (15):
- COHORT A= Amodiaquine + Artesunate (Active Comparator): Amodiaquine will be administered orally at 10mg/kg daily for 3days. Artesunate 50mg will be administered orally daily for 3days.For subjects >6months< 1 years 4mg/kg daily for 3 days
  Interventions: Drug: Amodiaquine + Artesunate
- cohort B= Lumefantrine +Artemether (Active Comparator): Artemether 20mg/Lumefantrine 120mg fixed combination administered daily for 3 days
  Interventions: Drug: Lumefantrine + Artemether
- cohort C = Artesunate + vitamin A (Experimental): Artesunate 50mg daily for 4days. if >6 months< 1 year 4mg/kg daily for 4days + Vitamin A 5000IU daily for 4days if < 1 year and 10,000IU daily for 4days if > 1 year respectively
  Interventions: Dietary Supplement: Artesunate + vitamin A
- Artesunate, vitamin E oral administration (Experimental): Artesunate 50mg daily for 4 days.if >6 months< 1 year 4mg/kg daily for 4 days + vitamin E 100mg daily administered orally to the experimental group 4 days.
  Interventions: Dietary Supplement: Artesunate + vitamin E
- cohort E will be given Artesunate and Zinc orally (Experimental): cohort E will be given Artesunate 50mg daily for 4 days. if > 6 months< 1 year 4mg/kg daily for 4 days + zinc gluconate 50mg orally daily for 4 days. if < 1 year 25 mg daily for 4 days
  Interventions: Dietary Supplement: Artesunate + Zinc
- cohort F= Artesunate and selenium will be given orally (Experimental): Artesunate 50mg daily for 4 days. if > 6 months< 1 year 4mg/kg daily for 4 days + selenium 100ug daily for 4 days. if < 1 year 50ug daily for 4 days.
  Interventions: Dietary Supplement: Artesunate + selenium
- cohort G = Amodiaqiune and Vitamin A will be given orally (Experimental): Amodiaquine 10mg/kg daily for 3 days + vitamin A 5000iu daily for 4 days if < 1 year. 10,000 IU daily for 4 days if > 1 year.
  Interventions: Dietary Supplement: Amodiaquine + vitamin A
- cohort H = amodiaquine and vitamin E administerd orally (Experimental): Amodiaquine 10mg/kg daily for 4 days + vitamin E 100 mg daily for 4 days
  Interventions: Dietary Supplement: Amodiaquine + Vitamin E
- cohort I = Amodiaquine and Zinc will be given orally (Experimental): Amodiaquine 10mg/kg daily for 4 days + zinc 50mg daily 4 days. if < 1 year 25 mg daily for 4 days.
  Interventions: Dietary Supplement: Amodiaquine + Zinc
- Cohort J = amodiaquine and selenium will be given orally (Experimental): Amodiaquine 10mg/kg daily for 4 days + selenium 100ug daily for 4 days if > 1 year. 50ug daily for 4 days if < 1 year.
  Interventions: Dietary Supplement: Amodiaquine + Selenium
- K= Artesunate+ vitamin A + vitamin E (Experimental): Tab Artesunate 50mg orally dly x 4 days + Vitamin A, 5000IU orally, dly x 4 days if ≤ 1yr. 10,000IU orally dly x 4days if > 1 yr + vitamin E 100 mg orally dly for 4 days
  Interventions: Dietary Supplement: Artesunate + vitamin A + vitamin E
- L = Artesunate+ Vitamin A + Zinc (Experimental): Tab Artesunate 50 mg daily for 4 days. Vitamin A 5OOOIU daily for 4 days if < 1 year. 10,000IU daily for 4 days if > 1 year. All administered orally.
  Interventions: Dietary Supplement: Artesunate + Vitamin A + Zinc
- M = Artesunate+ Vitamin A + selenium (Experimental): Artesunate 50 mg orally, daily for 4 days. Vitamin A 5000IU orally daily for 4 days if < 1 year. 10,000IU orally daily for 4 days if > 1 year.
  Interventions: Dietary Supplement: Artesunate + Vitamin A + Selenium
- N = Artesunate + Vitamin E + Zinc (Experimental): Artesunate 50mg daily for 4 days. vitamin E 100mg daily for 4 days. Zinc 50 mg daily for 4 days if > 1 year. 25 mg daily for 4 days if < 1 year.
  Interventions: Dietary Supplement: Artesunate + Vitamin E + Zinc
- O = Artesunate+ Vitamin E + Selenium (Experimental): Tab Artesunate 50 mg orally daily for 4 days. Vitamin E 100 mg orally daily for 4 days. Tab selenium 100 ug orally daily for 4 days if > 1 year. 50 ug orally daily for 4 days if < 1 year.
  Interventions: Dietary Supplement: Artesunate + Vitamin E + Selenium

INTERVENTIONS:
Drug: Amodiaquine + Artesunate — Intervention:the intervention in this group involves the use of standard antimalarial therapy for uncomplicated malaria based on WHO recommendation. artemisin based combination therapy will be used. amodiaquine will be administered via the oral route at a dose of 10mg/kg daily while artesunate will be administered orally at Artesunate 100mg stat, 50mg 8hrs later and 50mg bd x 3days
  Arms: COHORT A= Amodiaquine + Artesunate
Drug: Amodiaquine + Artesunate — Intervention:the intervention in this group involves the use of standard antimalarial therapy for uncomplicated malaria based on WHO recommendation. artemisinin based combination therapy will be used. amodiaquine will be administered via the oral route at a dose of 10mg/kg daily while artesunate will be administered orally at 100mg stat, 5omg 8hrs later and 50mg 12hrly for 3 days
  Arms: COHORT A= Amodiaquine + Artesunate
Drug: Lumefantrine + Artemether — Lumefantrine and artemether combination will be administered orally at a dose of 120/20mg daily for 3days
  Arms: cohort B= Lumefantrine +Artemether
Dietary Supplement: Artesunate + vitamin A — Artesunate will be administered orally at a dose of 100mg stat then 50 mg 8hrs later and 50mg 12hrly for 3days. vitamin A will be administered orally at a dose of 2000IU daily for 3 days
  Arms: cohort C = Artesunate + vitamin A
Dietary Supplement: Artesunate + vitamin E — Artesunate will be administered orally at 100mg stat, then 50mg 8hrs after and 50mg 12hrly for 3 days. Vitamin E will be administered orally at 100mg dly for 3 days.
  Arms: Artesunate, vitamin E oral administration
Dietary Supplement: Artesunate + Zinc — Artesunate will be administered orally at a dose of 100mg stat then 50mg 8hrs after and 50mg 12mg 12hrly for 3 days. Zinc gluconate will be administered orally at a dose of 50mg dly for 4 days
  Arms: cohort E will be given Artesunate and Zinc orally
Dietary Supplement: Artesunate + selenium — Artesunate will be administered orally at 100mg stat and 8hrs later 50mg. then 50mg 12hrly for 3 days. selenium will be administered orally at a dose of 100ug dly for 4 days
  Arms: cohort F= Artesunate and selenium will be given orally
Dietary Supplement: Amodiaquine + vitamin A — Amodiaquine will be administered orally at a dose of 10mg/kg dly for 3days. Vitamin A will be administered orally dly at a dose of 2000IU for 4 days
  Arms: cohort G = Amodiaqiune and Vitamin A will be given orally
Dietary Supplement: Amodiaquine + Vitamin E — Amodiaquine will be administered orally at a dose of 10mg/kg dly for 3days. vitamin E will be administered orally at a dose 100mg daily for 4 days
  Arms: cohort H = amodiaquine and vitamin E administerd orally
Dietary Supplement: Amodiaquine + Zinc — Amodiaquine will be administered orally at a dose of 10mg/kg dly for 3days. Zinc gluconate will be administered orally at a dose of 50mg dly for 4 days.
  Arms: cohort I = Amodiaquine and Zinc will be given orally
Dietary Supplement: Amodiaquine + Selenium — Amodiaquine will be administered orally at a dose of 10mg/kg daily for 3days. Selenium will be administered orally at a dose of 100ug daily for 4 days if > 1year. 50ug daily for 4 days if < 1 year.
  Arms: Cohort J = amodiaquine and selenium will be given orally
Dietary Supplement: Artesunate + vitamin A + vitamin E — Tab Artesunate 50mg orally daily for 4 days. Vitamin A, 5000IU orally daily for 4days if < 1 year. 10,000 IU orally daily for 4 days if > 1 year.
  Arms: K= Artesunate+ vitamin A + vitamin E
Dietary Supplement: Artesunate + Vitamin A + Zinc — Tab Artesunate 50 mg daily for 4 days. Vitamin A 5OOOIU daily for 4 days if < 1 year. 10,000IU daily for 4 days if > 1 year. All administered orally.
  Arms: L = Artesunate+ Vitamin A + Zinc
Dietary Supplement: Artesunate + Vitamin A + Selenium — Tab Artesunate 50 mg orally, daily for 4 days. Vitamin A 5000IU orally daily for 4 days if < 1 year. 10,000IU orally daily for 4 days if > 1 year.
  Arms: M = Artesunate+ Vitamin A + selenium
Dietary Supplement: Artesunate + Vitamin E + Selenium — Tab Artesunate 50 mg orally daily for 4 days. Vitamin E 100 mg orally daily for 4 days. Tab selenium 100 ug orally daily for 4 days if > 1 year. 50 ug orally daily for 4 days if < 1 year.
  Arms: O = Artesunate+ Vitamin E + Selenium
Dietary Supplement: Artesunate + Vitamin E + Zinc — Tab Artesunate administered orally at 50 mg daily for 4 days. Vitamin E 100 mg orally daily for 4 days. Tab Zinc 50 mg orally daily for 4 days if < 1 year. 25 mg orally daily for 4 days if > 1 year.
  Arms: N = Artesunate + Vitamin E + Zinc

SUMMARY:
In the last decade, the prevalence of malaria has been escalating at an alarming rate, especially in Africa. An estimated 300 to 500 million cases each year cause 1.5 to 2.7 million deaths, more than 90% occur in children under 5 years of age in Africa (WHO 1995). Malaria is Africa's leading cause of under-five mortality (20%) and constitutes 10% of the continent's overall disease burden. It accounts for 40% of public health expenditure, 30-50% of inpatient admissions, and up to 50% of outpatient visits in areas with high malaria transmission. Antioxidant micronutrients have immunomodulatory role and may have suppressive activity.

DETAILED DESCRIPTION:
The pathogenesis of plasmodial infection hinges on intracellular invasion of host erythrocyte and hepatocyte with possible generation of free radicals that may contribute to cellular membrane damage. This will make uninfected erythrocyte and hepatocyte to be more susceptible to merozoite invasion. Zinc and Selenium has immunomodulatory properties. They enhance cell-mediated immune response in malaria infection. This may help to adequately suppress schizont maturation and inhibit the release of merozoites. However, it is possible that they have a direct chemosuppressive or blood schizonticidal effect. The following research questions emanated from this hypothesis;

1. Do the micronutrients in question have direct suppressive or schizonticidal effect?
2. Can they be used as short course therapy with standard antimalarials in uncomplicated malaria?
3. Is their effect enhanced when used in combination with each other or with standard antimalarials?
4. Do they have any prophylactic benefit?
5. Can their use alter the course of established malaria infection?

ELIGIBILITY:
Inclusion Criteria:

* age of < 5 years
* asexual parasitemia of between 1,000 and 100,000/µl
* acute manifestation of malaria (e.g., history of fever in the preceding 24 hours or a temperature of >37.5°C at baseline)
* body weight between 5 and 30 kg
* ability to tolerate oral therapy
* informed consent by the legal representative of the subject (the parents, if possible), oral agreement of the child if appropriate
* resident in the study area for a duration of at least 4 weeks

Exclusion Criteria:

* adequate antimalarial treatment within the previous 7 days

  * use of micronutrients in the last 2 weeks
  * antibiotic treatment for a concurrent infection
  * hemoglobin level of <7 g/dl
  * hematocrit of <25%
  * leukocyte count of >15,000/µl
  * mixed plasmodial infection
  * severe malaria, any other severe underlying disease
  * concomitant disease masking assessment of the treatment response
  * inflammatory bowel disease, and any other disease causing fever

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
7-day cure rate | 4 weeks
  7-day Cure rate will be defined as initial and sustained parasite and symptom clearance with no increase in asexual parasitemia 48 h after the initiation of treatment and the absence of microscopically detected asexual parasitemia within 120 h of the commencement of treatment until day 7

SECONDARY OUTCOMES:
28-day cure rate. | 4 weeks
  the number of patients with clinical and parasitological cure by day 28 divided by the total number of patients who could be evaluated (per protocol population).

CONTACTS AND LOCATIONS:
Overall Officials: Osede Ignis Iribhogbe, MB.BS, M.Sc, Principal Investigator — Department of Pharmacology and Therapeutics, College of Medicine, Ambrose Alli University, Ekpoma; Ibrahim Oreagba, B.Pharm, M.Sc, Ph.D, Study Director — Deparment of Pharmacology, College of Medicine, University of Lagos, Nigeria; Elizabeth O. Agbaje, B.Sc, M.Sc, MPhil, Ph.D, Study Chair — Department of Pharmacology, College of Medicine University of Lagos, Nigeria; Prof. Onyebiguwa Patrick NMORSI, PhD, MD, Study Director — Dean, Faculty of Natural Sciences Ambrose Alli University Ekpoma
Locations (2):
- Nigeria (2):
  - Central Primary Health Centre, Ukpenu, Road, Ekpoma., Ekpoma, Edo
  - Faithdome Medical Centre, Ekpoma., Ekpoma, Esan West, Edo State

REFERENCES:
- [Background] Muller O, Becher H, van Zweeden AB, Ye Y, Diallo DA, Konate AT, Gbangou A, Kouyate B, Garenne M. Effect of zinc supplementation on malaria and other causes of morbidity in west African children: randomised double blind placebo controlled trial. BMJ. 2001 Jun 30;322(7302):1567. doi: 10.1136/bmj.322.7302.1567. PMID 11431296
- See also: chemoprophylactic effect of vitamin C in malaria — http://www.sciencealert.org